CLINICAL TRIAL: NCT05345730
Title: The Role of Left Atrial Fibrosis in Mitral Valve Repair Surgery (ALIVE Trial)
Acronym: ALIVE
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jolanda Kluin, Professor in Cardiothoracic Surgery, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL78497.018.21
Record Dates: First submitted 2022-01-12; First posted 2022-04-26 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Mitral Valve Disease; Mitral Regurgitation; Surgery; Cardiac Valve Disease; Mitral Valve Surgery; Mitral Valve Repair
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mitral valve insufficiency patients undergoing mitral valve repair surgery: The research population consists of mitral valve insufficiency patients scheduled for elective surgical mitral valve repair (N=20) according to the current European guideline criteria. These patients will undergo a cardiac MRI scan 2 weeks prior to surgery and 3 months after surgery.
  Interventions: Diagnostic Test: 3 DImensional Late Enhanced Gadolinium cardiac MRI scan

INTERVENTIONS:
Diagnostic Test: 3 DImensional Late Enhanced Gadolinium cardiac MRI scan — A cardiac MRI scan is made using late gadolinium enhancement to detect atrial fibrosis in the left atrium.

SUMMARY:
Rationale: Patients with mitral valve insufficiency suffer from left atrial remodeling. Atrial fibrosis is part of this remodeling process. The presence of atrial fibrosis is associated with adverse events.

Currently, mitral valve repair surgery is the ultimate treatment for severe primary mitral valve insufficiency. The main indications and timing for surgery are severe mitral valve insufficiency with symptoms or left ventricular dysfunction. However, the role of atrial fibrosis in this process remains undetermined despite its well-recognized clinical implications.

Characterization of atrial fibrosis patterns in mitral valve insufficiency patients might be potentially valuable for the indication and timing of mitral valve repair surgery in order to improve clinical outcomes.

To date, however, mitral valve insufficiency patients suffering from left atrial remodeling have hardly been studied using these new imaging techniques. Therefore, the investigators intend to combine advanced cardiac MRI and post-processing techniques prior to and after mitral valve repair surgery to gain more insight in the clinical implications of atrial fibrosis in this patient population.

It is hypothesized that the atrial fibrosis surface area paradoxically will increase after mitral valve surgery because of global shrinkage of the left atrium caused by the reversed remodeling process. As a consequence, more frequently atrial fibrosis related events including (paroxysmal) atrial fibrillation, may be observed in these patients.

Objective: To assess the effects of (reduced) volume overload on the left atrial wall texture (presence, amount and location of atrial fibrosis) and associated geometry and function in patients with mitral valve insufficiency, prior to and after mitral valve repair surgery.

Study design: Single center pilot study.

Study population: The research population consists of mitral valve insufficiency patients scheduled for elective surgical mitral valve repair (N=20) according to the current European guideline criteria.

DETAILED DESCRIPTION:
Patients with mitral valve insufficiency frequently suffer from left atrial remodeling, caused by volume overload and subsequent atrial dilatation. The associated myocardial stretch and increased wall tension, trigger a cascade of pathways leading to the occurrence of atrial fibrosis as part of the remodeling process. The clinical relevance of this atrial fibrosis, is that its presence is associated with an increased risk of atrial fibrillation, heart failure, pulmonary hypertension, a reduced quality of life and eventually a shorter life expectancy. In addition, in patients suffering from atrial fibrillation, the presence and amount of left atrial fibrosis was found to be a strong predictor for ablation efficacy and long-term outcome.

In daily clinical practice, mitral valve insufficiency is managed either by medical or surgical therapy. However, since medical therapy is often not sufficient for patients with severe primary mitral valve insufficiency, surgical intervention remains the ultimate treatment option for these patients. In general, valve repair is the preferred type of surgery, since it has better clinical results compared to valve replacement.

Currently, the indication and timing for valve surgery is mainly based on the severity of mitral valve insufficiency and the presence of symptoms and/or severity of left ventricular dysfunction. For clinical decision making and patient stratification for mitral valve surgery, the presence of atrial fibrosis is currently not taken in account, despite its well-recognized clinical implications.

Detection of atrial fibrosis patterns in patients with severe mitral valve insufficiency, however, may be potentially valuable for the indication and timing of mitral valve repair surgery to improve clinical outcomes. Improved insight into atrial fibrosis patterns and changes after mitral valve repair due to reverse remodeling, may help clinicians in their clinical decision making and timing for surgery.

Today, quantification of atrial fibrosis can be routinely performed using cardiac Magnetic Resonance Imaging (MRI) techniques and advanced post-processing tools, offering non-invasive tissue characterization in thin-walled structures.

To date, mitral valve insufficiency patients suffering from left atrial remodeling have hardly been studied using these new imaging techniques. Therefore, in this study, the investigators want to combine advanced cardiac MRI and post-processing techniques prior to and after mitral valve repair surgery to gain insight on the clinical role and predictive value of atrial fibrosis in this patient population.

In addition, the investigators aim to assess the effects of (reduced) volume overload on atrial wall texture, geometry and function.

It is hypothesized that the atrial fibrosis surface area paradoxically will increase after mitral valve surgery because of global shrinkage of the left atrium caused by the reversed remodeling process. As a consequence, more frequently atrial fibrosis related events including (paroxysmal) atrial fibrillation, may be observed in these patients.

With this insight, cardiac MRI can become clinical valuable for the indication and timing of surgical intervention in these patients. Surgical therapy might be renounced for example when a substantial increase of fibrosis surface is expected post-surgically causing a higher risk for atrial fibrillation, heart failure, pulmonary hypertension and a reduced quality of life. On the contrary, surgical therapy might be considered in an earlier stage of disease when the amount of fibrosis is still limited regarding its expected post-surgical development.

ELIGIBILITY:
Inclusion Criteria:

* Patients that meet the criteria for elective mitral valve repair surgery according to the European clinical guidelines (class I recommendation);

  * Symptomatic, chronic severe mitral valve insufficiency due to degenerative valve disease with a left ventricular ejection fraction >30%.
  * Asymptomatic, chronic severe mitral valve insufficiency due to degenerative valve disease with a left ventricular ejection fraction <60% and/or a left ventricular end-systolic diameter >45 mm.

Exclusion Criteria:

* not able to provide written informed consent.
* under the age of 18.
* with a history of cardiac surgery
* with atrial fibrillation
* with any comorbidity besides mitral valve insufficiency.
* with claustrophobia or any other contra-indication for magnetic resonance imaging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mitral valve insufficiency eligible for elective mitral valve repair surgery.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Severity of mitral valve insufficiency prior to surgery (regurgitation volume on MRI) | 2 weeks before surgery
  Severity of mitral valve insufficiency prior to surgery (defined as regurgitation volume in ml calculated using difference between left ventricular stroke volume (LVSV) and forward flow)
Severity of mitral valve insufficiency after surgery (regurgitation volume on MRI) | 3 months after surgery
  Severity of mitral valve insufficiency after surgery (defined as regurgitation volume in ml calculated using difference between left ventricular stroke volume (LVSV) and forward flow)
Left atrial remodelling prior to surgery (left atrial volume on MRI) | 2 weeks before surgery
  Left atrial volume (ml) measured by multislice volumetric method on MRI
Left atrial remodelling after surgery (left atrial volume on MRI) | 3 months after surgery
  Left atrial volume (ml) measured by multislice volumetric method on MRI
Left atrial remodelling prior to surgery (left atrial sphericity on MRI) | 2 weeks before surgery
  Calculated left atrial sphericity by using ratio of transverse and longitudinal diameters of the left atrium
Left atrial remodelling after surgery (left atrial sphericity on MRI) | 3 months after surgery
  Calculated left atrial sphericity by using ratio of transverse and longitudinal diameters of the left atrium
Left atrial remodelling prior to surgery (estimated wall tension) | 2 weeks before surgery
  Estimated wall tension using a calculation combining left atrial wall thickness, left atrial radius and pulmonary wedge pressure. Wall thickness and radius will be measured on MRI. Pulmonary wedge pressure will be measured by using a Swan-Ganz catheter during surgery
Left atrial remodelling after surgery (estimated wall tension) | 3 months after surgery
  Estimated wall tension using a calculation combining left atrial wall thickness, left atrial radius and pulmonary wedge pressure. Wall thickness and radius will be measured on MRI. Pulmonary wedge pressure will be measured by using a Swan-Ganz catheter during surgery
Presence and distribution patterns of LA fibrosis prior to surgery (quantification of fibrosis surface) | 2 weeks before surgery
  Quantification of fibrosis surface will be assessed by using dedicated software Cricle ADAS which is able to segment the left atrial wall and recognize fibrotic tissue by means of late gadolinium enhancement
Presence and distribution patterns of LA fibrosis after surgery (quantification of fibrosis surface) | 3 months after surgery
  Quantification of fibrosis surface will be assessed by using dedicated software Cricle ADAS which is able to segment the left atrial wall and recognize fibrotic tissue by means of late gadolinium enhancement
Presence and distribution patterns of LA fibrosis prior to surgery (geometric distribution of fibrosis) | 2 weeks before surgery
  Geometric distribution of fibrosis in the left atrium will be assessed using dedicated software Circle ADAS. The software is able to segment the left atrial and define the three-dimensional geometric distribution of fibrotic tissue
Presence and distribution patterns of LA fibrosis after surgery (geometric distribution of fibrosis) | 3 months after surgery
  Geometric distribution of fibrosis in the left atrium will be assessed using dedicated software Circle ADAS. The software is able to segment the left atrial and define the three-dimensional geometric distribution of fibrotic tissue
Blood flow patterns in the left atrium prior to surgery (flow velocity) | 2 weeks before surgery
  Blood flow patterns in the left atrium will be assessed by measuring flow velocity using synthetic velocity fields as well as Poiseuille flow. This will be done with dedicated software Circle
Blood flow patterns in the left atrium after surgery (flow velocity) | 3 months after surgery
  Blood flow patterns in the left atrium will be assessed by measuring flow velocity using synthetic velocity fields as well as Poiseuille flow. This will be done with dedicated software Circle
Blood flow patterns in the left atrium prior to surgery (kinetic energy) | 2 weeks before surgery
  Kinetic energy of the blood flow patterns will be measured by using dedicated software Circle by means of advanced 4D flow CRM techniques defining global kinetic energy
Blood flow patterns in the left atrium after surgery (kinetic energy) | 3 months after surgery
  Kinetic energy of the blood flow patterns will be measured by using dedicated software Circle by means of advanced 4D flow CRM techniques defining global kinetic energy

SECONDARY OUTCOMES:
Change of fibrosis associated biomarkers derived from blood samples (prior to surgery versus after surgery) - NT-proBNP | 2 weeks before surgery and 3 months after surgery
  NT-proBNP
Change of fibrosis associated biomarkers derived from blood samples (prior to surgery versus after surgery) - TGF-β | 2 weeks before surgery and 3 months after surgery
  TGF-β
Change of fibrosis associated biomarkers derived from blood samples (prior to surgery versus after surgery) - TNF-alfa | 2 weeks before surgery and 3 months after surgery
  TNF-alfa
Change of fibrosis associated biomarkers derived from blood samples (prior to surgery versus after surgery) - Galectin-3 | 2 weeks before surgery and 3 months after surgery
  Galectin-3
Change of fibrosis associated biomarkers derived from blood samples (prior to surgery versus after surgery) - MMS | 2 weeks before surgery and 3 months after surgery
  MMS
Change of fibrosis associated biomarkers derived from blood samples (prior to surgery versus after surgery) - Angiotensin II | 2 weeks before surgery and 3 months after surgery
  Angiotensin II

CONTACTS AND LOCATIONS:
Overall Officials: Jolanda Kluin, M.D., PhD, Principal Investigator — j.kluin@amsterdamumc.nl
Locations (1):
- AmsterdamUMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
When asked for, a construction will be made to share data. At the end of the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT05345730/Prot_SAP_000.pdf